CLINICAL TRIAL: NCT05971706
Title: Impact of Ozone Application in Periodontitis Patients
Brief Title: Ozone Application in Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Principle Investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ozone
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Periodontitis
Keywords: periodontitis; ozone; treatment
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone (Experimental): Gaseous ozone was applied immediately after non-surgical periodontal treatment
  Interventions: Device: Ozone therapy using a device (Ozone DTA Ozone Generator, Denta Tec Dental AS, Norway); Procedure: Non-surgical periodontal treatment
- control (Active Comparator): Only non-surgical periodontal treatment was applied
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Device: Ozone therapy using a device (Ozone DTA Ozone Generator, Denta Tec Dental AS, Norway) — Ozone therapy procedures will be performed immediately after non-surgical periodontal treatment and three times (every third day) within one week using a device equipped with a periodontal tip according to equipment producer recommendations. The periodontal tip will be halted 1 mm short of the pocket depth. Ozone will be applied only to the pockets; which depth is equal to or greater than 5 mm. Ozone application time to the pockets will be 30 seconds at a fixed concentration of 2,100 ppm (80% oxygen) through a connected handpiece.
  Arms: ozone
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal treatment consists of oral hygiene instructions, full mouth supragingival scaling using hand instruments, ultrasonic devices, polishing, and subgingival debridement under local anesthesia with sharp Gracey and Universal curettes and ultrasonic instruments in a single appointment.

SUMMARY:
This clinical trial aims to evaluate the clinical, biochemical and microbiological efficacy of ozone treatment as an adjunct to nonsurgical periodontal treatment (NSPT) in periodontitis patients. The main question it aims to answer is:

• Is the application of gaseous ozone, as an adjunct to NSPT, to periodontal pockets in patients with periodontitis alters the clinical periodontal parameters, gingival crevicular fluid levels of inflammatory cytokines, and periodontal pathogens compared to NSPT alone? The study will be performed according to a split-mouth design, the contralateral quadrants with similar periodontal status in each patient will be randomly allocated to one of the following two different treatment modalities.

Participants will be applied NSPT consisting of supra and subgingival debridement.

* NSPT will be applied alone in one quadrant
* In addition to NSPT, ozone therapy procedures were performed using a device at contralateral sites.

Researchers will compare the sites with and without ozone therapy in addition to NSPT to see if ozone therapy adjunct to the NSPT affects clinical, biochemical, and microbiological changes

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* no periodontal treatment within 6 months from the enrollment date
* no antibiotics or anti-inflammatory medication taken within 6 months from the enrollment date
* no smokers
* no pregnancy or lactation at the time of the stud
* no contraindication for periodontal treatment and ozone application

Exclusion Criteria:

* Participants will be excluded if they had less than 20 teeth, partial dentures, or fixed prosthodontics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline (prior to therapy)
  Probing pocket depth: The distance from the base of the pocket to the gingival margin. Measurements will be made at six points on all teeth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing pocket depth | 3rd month after treatment
  robing pocket depth: The distance from the base of the pocket to the gingival margin. Measurements will be made at six points on all teeth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.

SECONDARY OUTCOMES:
Plaque index (Silness & Löe, 1964) | Baseline (prior to therapy)
  Plaque index (Silness & Löe, 1964):
  0: Absence of microbial plaque
  1. Thin plaque layer at the gingival margin, only detectable by scraping with a probe
  2. Moderate layer of plaque in the along the gingival margin; interdental spaces free, but plaque is visible to naked eye
  3. Abundant plaque along with the gingival margin; interdental places filled with plaque
Plaque index (Silness & Löe, 1964) | 3rd month
  Plaque index (Silness & Löe, 1964):
  0: Absence of microbial plaque
  1. Thin plaque layer at the gingival margin, only detectable by scraping with a probe
  2. Moderate layer of plaque in the along the gingival margin; interdental spaces free, but plaque is visible to naked eye
  3. Abundant plaque along with the gingival margin; interdental places filled with plaque
Gingival Index ( Löe & Silness,1963) | Baseline (prior to therapy)
  0 = normal gingiva
  1. = mild inflammation - slight change in color and slight edema but no bleeding on probing
  2. = moderate inflammation - redness, edema and glazing, bleeding on probing
  3. = severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index ( Löe & Silness,1963) | 3rd month
  0 = normal gingiva
  1. = mild inflammation - slight change in color and slight edema but no bleeding on probing
  2. = moderate inflammation - redness, edema and glazing, bleeding on probing
  3. = severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Bleeding on probing | Baseline (prior to therapy)
  A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth (Ainamo & Bay 1975).
Bleeding on probing | 3rd month
  A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth (Ainamo & Bay 1975).
Proportions of bacterial species | Baseline (prior to therapy)
  Subgingival plaque sampling will be performed at the 3 deepest pockets with a probing depth equal to or higher than 5mm in each treatment site with no endodontic or furcation involvement using 2 standardized sterile paper points. One will be inserted at a 45-degree angle and the other will be inserted parallel to the tooth axis and left in place for 30 seconds. Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia will be evaluated.
Proportions of bacterial species | 1st month
  Subgingival plaque sampling will be performed at the 3 deepest pockets with a probing depth equal to or higher than 5mm in each treatment site with no endodontic or furcation involvement using 2 standardized sterile paper points. One will be inserted at a 45-degree angle and the other will be inserted parallel to the tooth axis and left in place for 30 seconds. Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia will be evaluated.
Proportions of bacterial species | 3rd month
  Subgingival plaque sampling will be performed at the 3 deepest pockets with a probing depth equal to or higher than 5mm in each treatment site with no endodontic or furcation involvement using 2 standardized sterile paper points. One will be inserted at a 45-degree angle and the other will be inserted parallel to the tooth axis and left in place for 30 seconds. Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia will be evaluated.
Inflammatory parameter levels in gingival crevicular fluid | Baseline (prior to therapy)
  Subgingival plaque sampling will be performed at the 3 deepest pockets with a probing depth equal to or higher than 5mm in each treatment site with no endodontic or furcation involvement using sterile paper strips. Gingival crevicular fluid Tumor necrotizing factor-alpha, interleukin-1beta, interleukin-6, interleukin-8 levels will be evaluated.
Inflammatory parameter levels in gingival crevicular fluid | 1st month
  Subgingival plaque sampling will be performed at the 3 deepest pockets with a probing depth equal to or higher than 5mm in each treatment site with no endodontic or furcation involvement using sterile paper strips. Gingival crevicular fluid Tumor necrotizing factor-alpha, interleukin-1beta, interleukin-6, interleukin-8 levels will be evaluated.
Inflammatory parameter levels in gingival crevicular fluid | 3rd month
  Subgingival plaque sampling will be performed at the 3 deepest pockets with a probing depth equal to or higher than 5mm in each treatment site with no endodontic or furcation involvement using sterile paper strips. Gingival crevicular fluid Tumor necrotizing factor-alpha, interleukin-1beta, interleukin-6, interleukin-8 levels will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No